CLINICAL TRIAL: NCT05371171
Title: Management of Skin Graft Donor Site Wound in Aged Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201801010
Record Dates: First submitted 2022-02-24; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-02

CONDITIONS: Skin Regrafting; Donor Site of Skin Grafting; Vancouver Scar Scale
MeSH Terms: interventions — Skin Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin graft (Experimental)
  Interventions: Procedure: skin graft
- no skin graft (Placebo Comparator)
  Interventions: Procedure: no skin graft

INTERVENTIONS:
Procedure: skin graft — In the experimental group, the operative plan was to consider taking a 15% larger amount than necessary and replace over-harvested skin back onto the donor site in an island manner. Any remaining skin graft was returned to the donor site and a polyurethane dressing [Alleyvn, Smith, & Nephew] was placed on the regrafted skin for fixation
  Arms: skin graft
Procedure: no skin graft — In the experimental group, the operative plan was to consider taking a 15% larger amount than necessary and replace over-harvested skin back onto the donor site in an island manner. Any remaining skin graft was returned to the donor site and a polyurethane dressing [Alleyvn, Smith, & Nephew] was placed on the regrafted skin for fixation
  Arms: no skin graft

SUMMARY:
The complication of donor site in skin grafting often acts as a causing factor for extended treatment period. The elderly individuals tend to be afflicted by impaired wound healing. Herein, the investigators presented the outcome of skin regrafting in the elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patient who need to perform skin grafting surgery

Exclusion Criteria:

1. All patient who cannot be half or general anesthetized
2. severe comorbidities

Ages: 60 Months to 99 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
healing time | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Wan Fang Hospital, Taipei County, Taiwan